CLINICAL TRIAL: NCT03608904
Title: A Quantitative Connectivity Assessment of Music Listening Compared to Spoken Word in Ischemic Stroke Recovery, as Measured by Functional MRI (fMRI).
Brief Title: Stroke Recovery and Music or No Music
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Methodist Hospital Research Institute (Other)
Collaborators: Houston Methodist Centers of Performing Arts Medicine (Unknown)
Responsible Party: Principal Investigator, John J. Volpi, MD, Principal Investigator, Neurologist, The Methodist Hospital Research Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Pro00015563
Record Dates: First submitted 2018-04-13; First posted 2018-08-01 (Actual); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Ischemic Stroke
Keywords: Stroke; Music; Ischemic Stroke; fMRI; functional MRI
MeSH Terms: conditions — Ischemic Stroke; Stroke | interventions — Auditory Perception

STUDY DESIGN:
Intervention Model Description: Participants will be exposed to music or no music (spoken words only) during their fMRI scans.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music Listening (Experimental): Familiar and unfamiliar music selections, listening duration of approximately 15 minutes, three times daily, 90-day listening duration.
  Interventions: Other: Music listening
- Spoken word (language) listening (Placebo Comparator): Familiar and unfamiliar spoken word (language) selections, listening duration of approximately 15 minutes, three times daily, 90-day listening duration.
  Interventions: Other: Spoken word (language) listening

INTERVENTIONS:
Other: Music listening — Familiar and unfamiliar music selections, listening duration of approximately 15 minutes, three times daily, 90-day listening duration.
  Arms: Music Listening
Other: Spoken word (language) listening — Familiar and unfamiliar spoken word (language) selections, listening duration of approximately 15 minutes, three times daily, 90-day listening duration.
  Arms: Spoken word (language) listening

SUMMARY:
The primary outcome of this study is to determine the quantitative increase in connectivity, as measured by fMRI brain and calculated as a percent increase from baseline in patients with ischemic stroke. Eligible patients will receive a listening session of music or spoken word listening, 30 days to 5 years following ischemic stroke. Assessments will include modified Rankin Scale, National Institute of Health Stroke Scale, functional Magnetic Resonance Imaging, motor function tests, and neuropsychological evaluations. Assessments occur at baseline, day 45, and day 90 after starting listening sessions.

DETAILED DESCRIPTION:
This is a prospective, investigator-blinded and outcome assessor-blinded, randomized, single-center study in subjects 18-90 years old who have sustained an ischemic stroke within 30 days to 5 years. Study subjects will be randomized 1:1 to receive one of two types of listening sessions: music or spoken word (language) listening. Each arm will enroll a total of ten subjects, with a total study population of 20 subjects. Subjects will follow a 90-day listening schedule.

Subjects will complete a baseline Montreal Cognitive Assessment (MoCA), National Institute of Health Stroke Scale (NIHSS), modified Rankin Score (mRS), motor function tests, neuropsychological evaluations and functional magnetic resonance imaging (fMRI) brain evaluation. Follow-up evaluations on day 45 (+/- 7 days) and on day 90 (+/-7days) and will include NIHSS/mRS, motor function tests, neuropsychological evaluations and fMRI Brain evaluation.

All subjects will continue to receive standard of care treatment for stroke as directed by their physician(s) regardless of study enrollment.

The primary objective is to determine the quantitative increase in connectivity, as measured by fMRI brain and calculated as a percent increase from baseline.

The secondary objectives include the effect of music and language listening in improving motor function and neuropsychological development in patients with an ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

1. Ischemic Stroke 30 days to 5 years days prior to enrollment
2. Age 18-90
3. Modified Rankin Score (mRS) 1-3, inclusive, post-qualifying event (for a history of multiple strokes, baseline mRS is 0-1 AND a lower value than the qualifying mRS)
4. A measureable deficit either in motor or speech/cognition that can be assessed using standardized testing
5. Fluency in English (written and verbal)
6. Demonstrates willingness to participate in study and complete all schedule of events

Exclusion Criteria:

1. Severe cognitive impairment, as determined by investigator using the baseline MoCA score
2. Comorbid neurological disease that may interfere with rehabilitation
3. Psychiatric disorder or taking psychoactive medication that may interfere with completing study
4. Inability to complete music listening exercises
5. Alcohol or drug abuse
6. Hearing impairment
7. Contraindication to scheduled fMRI Brain evaluations
8. Pregnant women

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-07-21 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Connectivity as Measured by Functional Magnetic Resonance Imaging (fMRI) at Baseline as Compared to Post-Listening Exposure at Days 45 and 90. | Change from Baseline to Days 45 and 90
  To determine quantitative increase in connectivity of music and/or spoken word (language) listening, as measured by fMRI brain, and calculated as a percent increase from baseline.

SECONDARY OUTCOMES:
Change in Motor Function Test Pinch Grip (pounds) at Baseline as Compared to Post-Listening Exposure at Day 45 and Day 90. | Change from Baseline to Days 45 and 90
  To assess the effect of music and/or spoken word (language) listening in improving motor function test of pinch grip.
Change in Motor Function Test Grip Strength (pounds) at Baseline as Compared to Post-Listening Exposure at Days 45 and 90. | Change from Baseline to Days 45 and 90
  To assess the effect of music and/or spoken word (language) listening in improving motor function test of grip strength.
Change in Grooved Pegboard Test (seconds) at Baseline as Compared to Post-Listening Exposure at Days 45 and 90. | Change from Baseline to Days 45 and 90
  To assess the effect of music and/or spoken word (language) listening in improving motor function test of grooved pegboard test.
Change in Action Research Arm Test (score) at Baseline as Compared to Post-Listening Exposure at Days 45 and 90. | Change from Baseline to Days 45 and 90
  To assess the effect of music and/or spoken word (language) listening in improving motor function test of Action Research Arm Test (ARAT).
Change in Timed Up and Go (seconds) at Baseline as Compared to Post-Listening Exposure at Days 45 and 90. | Change from Baseline to Days 45 and 90
  To assess the effect of music and/or spoken word (language) listening in improving motor function test of Timed Up and Go.
Change in 10 Meter Walk Test (seconds) at Baseline as Compared to Post-Listening Exposure at Days 45 and 90. | Change from Baseline to Days 45 and 90
  To assess the effect of music and/or spoken word (language) listening in improving motor function test of 10 meter walk test.
Change in Modified Rankin Score (score) at Baseline as Compared to Post-Listening Exposure at Days 45 and 90. | Change from Baseline to Days 45 and 90
  To assess the effect of music and/or spoken word (language) listening in improvement of disability score.
Change in National Institutes of Health Stroke Scale (score) at Baseline as Compared to Post-Listening Exposure at Days 45 and 90. | Change from Baseline to Days 45 and 90
  To assess the effect of music and/or spoken word (language) listening in improvement of standardized stroke score.
Change in Neuropsychological Evaluation Wechsler Adult Intelligence Scale-IV: Digit Span (score) at Baseline as Compared to Post-Listening Exposure at Days 45 and 90. | Change from Baseline to Days 45 and 90
  To assess the effect of music and/or spoken word (language) listening in improvements of neuropsychology evaluation of an aural test of immediate attention and working memory.
Change in Neuropsychological Evaluation Albert's Test (score) at Baseline as Compared to Post-Listening Exposure at Days 45 and 90. | Change from Baseline to Days 45 and 90
  To assess the effect of music and/or spoken word (language) listening in improvement of neuropsychology evaluation of a line cancellation test of visual attention/neglect.
Change in Neuropsychological Evaluation Rey Complex Figure Test and Recognition Trial (score) at Baseline as Compared to Post-Listening Exposure at Days 45 and 90. | Change from Baseline to Days 45 and 90
  To assess the effect of music and/or spoken word (language) listening in improvement of neuropsychology evaluation of a drawing test used to assess planning, organization and visual-spatial skills.
Change in Neuropsychological Evaluation MAST (score) at Baseline as Compared to Post-Listening Exposure at Days 45 and 90. | Change from Baseline to Days 45 and 90
  To assess the effect of music and/or spoken word (language) listening in improvement of neuropsychology evaluation of a language measure for patients with aphasia.
Change in Neuropsychological Evaluation MAE Token Test (score) at Baseline as Compared to Post-Listening Exposure at Days 45 and 90. | Change from Baseline to Days 45 and 90
  To assess the effect of music and/or spoken word (language) listening in improvement of neuropsychology evaluation of an aural language comprehension measure.
Change in Neuropsychological Evaluation Boston Naming Test (score) at Baseline as Compared to Post-Listening Exposure at Days 45 and 90. | Change from Baseline to Days 45 and 90
  To assess the effect of music and/or spoken word (language) listening in improvement of neuropsychology evaluation of a test of confrontation naming.
Change in Neuropsychological Evaluation Phonemic Fluency (score) at Baseline as Compared to Post-Listening Exposure at Days 45 and 90. | Change from Baseline to Days 45 and 90
  To assess the effect of music and/or spoken word (language) listening in improvement of neuropsychology evaluation of a generative naming test.
Change in Neuropsychological Evaluation Semantic fluency (score) at Baseline as Compared to Post-Listening Exposure at Days 45 and 90. | Change from Baseline to Days 45 and 90
  To assess the effect of music and/or spoken word (language) listening in improvement of neuropsychology evaluation of a generative naming test.
Change in Neuropsychological Evaluation Wide Range Achievement Test-4 Reading (score) at Baseline as Compared to Post-Listening Exposure at Days 45 and 90. | Change from Baseline to Days 45 and 90
  To assess the effect of music and/or spoken word (language) listening in improvement of neuropsychology evaluation of a single-word reading measure that can be used, in some, to assess premorbid intellectual abilities.
Change in Neuropsychological Evaluation Trail Making Test-A (score) at Baseline as Compared to Post-Listening Exposure at Days 45 and 90. | Change from Baseline to Days 45 and 90
  To assess the effect of music and/or spoken word (language) listening in changes of a neuropsychology evaluation of a speeded psychomotor test of attention.
Change in Neuropsychological Evaluation Trail Making Test-B (score) at Baseline as Compared to Post-Listening Exposure at Days 45 and 90. | Change from Baseline to Days 45 and 90
  To assess the effect of music and/or spoken word (language) listening in improvement of neuropsychology evaluation of a speeded psychomotor test of alternating attention/working memory.
Change in Neuropsychological Evaluation Hopkins Verbal Learning Test-Revised (score) at Baseline as Compared to Post-Listening Exposure at Days 45 and 90. | Change from Baseline to Days 45 and 90
  To assess the effect of music and/or spoken word (language) listening in changes of a neuropsychology evaluation of a rote verbal learning and test.
Change in Neuropsychological Evaluation Brief Visuospatial Memory Test-Revised (score) at Baseline as Compared to Post-Listening Exposure at Days 45 and 90. | Change from Baseline to Days 45 and 90
  To assess the effect of music and/or spoken word (language) listening in improvement of neuropsychology evaluation of a visual learning and memory test.
Change in Neuropsychological Evaluation Clock Test (score) at Baseline as Compared to Post-Listening Exposure at Days 45 and 90. | Change from Baseline to Days 45 and 90
  To assess the effect of music and/or spoken word (language) listening in improvement of neuropsychology evaluation of a measure of conceptualization, planning, organization, and visual-spatial skills.
Change in Neuropsychological Evaluation Beck Depression Inventory-II (score) at Baseline as Compared to Post-Listening Exposure at Days 45 and 90. | Change from Baseline to Days 45 and 90
  To assess the effect of music and/or spoken word (language) listening in improvement of neuropsychology evaluation of a test to measure depression.
Change in Neuropsychological Evaluation Generalized Anxiety Disorder 7-item(score) at Baseline as Compared to Post-Listening Exposure at Days 45 and 90. | Change from Baseline to Days 45 and 90
  To assess the effect of music and/or spoken word (language) listening in improvement of neuropsychology evaluation of a test to measure generalized anxiety.
Change in Neuropsychological Evaluation The Stroke-Adapted Sickness Impact Profile (SA-SIP30) (score) at Baseline as Compared to Post-Listening Exposure at Days 45 and 90. | Change from Baseline to Days 45 and 90
  To assess the effect of music and/or spoken word (language) listening in improvement of neuropsychology evaluation of a post-stroke quality of life measure.

CONTACTS AND LOCATIONS:
Overall Officials: John J Volpi, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Houston Methodist, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
No plans at to share individual subject data at this time.

REFERENCES:
- [Background] Karmonik C, Brandt A, Anderson J, Brooks F, Lytle J, Silverman E, Frazier JT. Music Listening modulates Functional Connectivity and Information Flow in the Human Brain. Brain Connect. 2016 Oct;6(8):632-641. doi: 10.1089/brain.2016.0428. Epub 2016 Jul 27. PMID 27464741